CLINICAL TRIAL: NCT02000258
Title: Effect of Tunnel Placements on Clinical and MRI Findings Two Years After Anterior Cruciate Ligament Reconstruction With Double-Bundle Technique
Brief Title: Effect of Tunnel Placements on Clinical and MRI Findings Two Years After ACL Reconstruction With DB Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: R02071
Record Dates: First submitted 2013-10-30; First posted 2013-12-04 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-11

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: Anterior cruciate ligament reconstruction; Double-bundle; MRI; Graft location
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Double-bundle ACL reconstruction (Other): Double-bundle ACL reconstruction
  Interventions: Procedure: Double-bundle ACL reconstruction
- Magnetic resonance imaging (MRI) (Other): MRI of the ACL double-bundle reconstructed knee was done at 2 years after surgery.
  Interventions: Device: Magnetic resonance imaging (MRI)

INTERVENTIONS:
Procedure: Double-bundle ACL reconstruction
  Arms: Double-bundle ACL reconstruction
Device: Magnetic resonance imaging (MRI) — MRI sequences were as follows: sagittal T1-weighted, proton density (PD)-weighted and T2-weighted fast spin echo (FSE) images with 4 mm slice and 1 mm gap, coronal T1-weighted and fat-saturated T2-weighted FSE images with 4 mm slice and 1 mm gap, axial fat saturated PD FSE images with 4 mm slice and 1 mm gap and oblique sagittal and oblique coronal T1 FSE images along AM graft plane with 3 mm slice and 0.3 mm gap.
  Other Names: MRI evaluations were made with a 1.5-T Signa Excite HD imager (GE Healthcare, Milwaukee, WI) by use of an eight-channel receiver/transmitter extremity coil.; The interpretation of the images was made with the Impax DS 3000 workstation (Agfa HealthCare, Mortsel, Belgium)
  Arms: Magnetic resonance imaging (MRI)

SUMMARY:
Purpose: To find out whether the clinical and MRI findings two years after anterior cruciate ligament (ACL) reconstruction were associated with each other so that MRI-based graft invisibility in the anteromedial (AM) graft would have an impact on anteroposterior stability of the knee, and MRI-based posterolateral (PL) graft invisibility on rotational stability of the knee.

Methods: 75 patients. One experienced orthopaedic surgeon performed all double-bundle (DB) ACL reconstructions. Two independent examiners made the clinical examinations at the two-year follow-up: clinical examination of the knee, KT-1000, International Knee Documentation Committee (IKDC) and Lysholm knee evaluation scores and IKDC functional score. The MRI evaluations were made by two musculoskeletal radiologists separately and the means of these measurements were used.

ELIGIBILITY:
Inclusion Criteria:

* primary ACL reconstruction, closed growth plates

Exclusion Criteria:

* ligament injury to the opposite knee

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2003-03; Primary Completion 2010-09 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The location of the ACL grafts in the insertion site in the femur and in the tibia reported as percentages | 2 years after surgery
  The measurements of the graft location from the MRI were made by two musculoskeletal radiologists separately and the means of these measurements were used. In brief, first the centers of the tunnels were measured from sagittal images referring to the Blumensaat's line and to the posterior femoral condyle. Then these were divided with the maximum diameters of the femoral condyle parallel to and perpendicular to the Blumensaat's line. In the tibial side, the centers of the tunnels were measured from the anterior edge of the tibial plateau and then divided with the maximum diameter of the plateau, which was measured from the sagittal view.
The visibility of the ACL grafts measured from the MRI | 2 years after surgery
  Two musculoskeletal radiologists made the interpretation of the images separately and the means of these measurements were used. A graft was considered visible when intact graft fibers were seen. The graft was considered partially visible when only few graft fibers were seen. The graft was considered invisible when no graft fibers were seen.

SECONDARY OUTCOMES:
KT-1000 measurement (mm) of the knees of 61 patients | 2 years after surgery
  KT-1000 measurements were reported as millimeters.
International Knee Documentation Committee (IKDC) functional score | 2 years after surgery
  IKDC functional score was used to evaluate knee functions (IKDC scale: 0-10). Full function without any limitations was scored as 10, while zero indicated that those patients were unable to perform their daily activities.
Lysholm knee evaluation score | 2 years after surgery
  Patients completed the Lysholm knee score, which measures subjective functions e.g. squatting and running. The scale is 0-100, 100 being perfect functioning of the knee.
Clinical evaluation of the knees on the basis of International Knee Documentation Committee (IKDC) examination form | 2 years after surgery
  The clinical evaluation was performed on the basis of IKDC knee examination form, which gives the final score A-D. A being normal, B nearly normal, C abnormal and D severely abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: Timo Järvelä, MD, PhD, Study Chair — Arthroscopic and sports medicine center Omasairaala, Helsinki, Finland
Locations (1):
- Tampere University hospital, Tampere, Pirkanmaa, Finland